CLINICAL TRIAL: NCT03977740
Title: Efficacy of Chest PNF on Pulmonary Function in Patients With Parkinson's Diseases
Brief Title: Chest PNF on Pulmonary Function in Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Subhasish Chatterjee (Other)
Responsible Party: Sponsor-Investigator, Subhasish Chatterjee, clinical professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IEC-1111
Record Dates: First submitted 2019-05-27; First posted 2019-06-06 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chest PNF (Experimental): participants received conventional chest physiotherapy along with chest PNF technique 5 days for 1 week.
  Chest PNF technique includes oblique downward pressure at the sternum, diagonal pressure at lower rib cage at the supine line, caudal medial pressure at side lying, Caudal pressure at ribcage at prone lying, dorsal and caudal pressure at prone on the elbow.
  Interventions: Other: chest PNF
- Conventional (Active Comparator): participants received conventional chest physiotherapy treatment, which includes Deep breathing exercise, Diaphragmatic breathing exercise, segmental breathing exercise and purse lip breathing and incentive spirometer
  Interventions: Other: Conventional

INTERVENTIONS:
Other: chest PNF — Chest PNF technique includes oblique downward pressure at sternum, diagonal pressure at lower rib cage at supine line, caudal medial pressure at side lying, Caudal pressure at ribcage at prone lying, dorsal and caudal pressure at prone on elbow.
  Arms: chest PNF
Other: Conventional — conventional chest physiotherapy treatment, which includes Deep breathing exercise, Diaphragmatic breathing exercise, segmental breathing exercise and purse lip breathing and incentive spirometer
  Arms: Conventional

SUMMARY:
Background: Parkinson disease (PD) is a progressive neurodegenerative disorder and characterized by tremor, rigidity and bradykinesia. Almost 84% of PD patient develops respiratory abnormalities and pointed as the most common cause of death. Airway obstruction, trunk muscle rigidity is the common cause of respiratory abnormalities.

Purpose: The main purpose of the study will evaluate the efficacy of chest PNF on pulmonary function and chest wall mobility in PD.

Methods: 20 participants will be recruited for study purpose and divide into two groups. Group= A will be the control group and participants will receive conventional treatment which includes deep breathing exercise and segmental breathing exercise, incentive spirometry etc for one week. Group= B participants will receive chest PNF exercise along with conventional treatment for a week. Pretreatment and post-treatment data will be recorded by the help of PFT (FVC, FEV1 & FEV1/FVC) and chest wall expansion at axillary and xiphisternal level for data analysis. Data analysis will be done by paired t-test for within group and independent t-test will be used for the between-group variable. The level of significance will be set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Grade 3 to grade 5 Parkinson patients according to Hoehn Yahar scale
2. MMSE score >23.
3. Age 50-70 yrs.
4. Both Male and Female.

Exclusion Criteria:

1. Previous history of cardiac and pulmonary surgery.
2. History of flail chest.
3. Individual affected by neurological disorder other than PD.
4. Uncooperative patients.
5. Individual with the psychosomatic disorder.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-06-10 (Estimated); Study Completion 2019-06-10 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Function Test (PFT) | changes bwtween baseline to 1 week
  Pulmonary functions parameters FVC in litre, FEV1 in litre and ratio between FVC/FEV1 will be recorded with PFT

SECONDARY OUTCOMES:
chest wall expansion by inch tape | changes bwtween baseline to 1 week
  chest wall expansion will be measured at axillary and xiphisternal level

CONTACTS AND LOCATIONS:
Locations (1):
- MMIPR, Ambāla, Haryana, India

IPD SHARING:
Plan to Share IPD: No